CLINICAL TRIAL: NCT04202406
Title: Effect of Preoperative Acetaminophen-Codeine-Caffeine Combination on Inferior Alveolar Nerve Block Success in Patients With Symptomatic Irreversible Pulpitis: Randomized Double-blind Controlled Trial
Brief Title: Preoperative Acetaminophen- Caffeine- Codeine Combination and Anaesthetic Success in Patients With Acute Pulpitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Mohammed Abdallah Morsi, Post graduate student, Department of Endodontics, Faculty of Dentistry,Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CEBD-CU-2019-03-13
Record Dates: First submitted 2019-12-16; First posted 2019-12-17 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Symptomatic Irreversible Pulpitis
Keywords: Postoperative pain; Paracetamol; Placebo; Single visit root canal treatment
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen; Codeine; Caffeine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Acetaminophen, codeine,and caffeine (Experimental): Oral single dose of Combination of 1000mg acetaminophen- 16mg codeine- 60mg caffeine.
  Interventions: Drug: Acetaminophen and codeine and caffeine
- Acetaminophen (Experimental): Oral single dose of 1000mg acetaminophen.
  Interventions: Drug: Acetaminophen
- Placebo (Placebo Comparator): Maize starch.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetaminophen and codeine and caffeine — The patient will receive pretreatment oral single dose of Combination of 1000mg acetaminophen- 16mg codeine- 60mg caffeine 1 hour before treatment.
  Arms: Acetaminophen, codeine,and caffeine
Drug: Acetaminophen — The patient will receive pretreatment oral single dose of 1000mg acetaminophen alone 1 hour before treatment.
  Arms: Acetaminophen
Drug: Placebo — The patient will receive placebo (starch) 1hour before treatment.
  Arms: Placebo

SUMMARY:
The aim of the study is to evaluate the effect of preoperative administration of acetaminophen- codeine -caffeine combination on the success of the inferior alveolar nerve block versus bacetaminophen alone or placebo in patients with symptomatic irreversible pulpitis.

DETAILED DESCRIPTION:
After ensuring eligibility, patients will be given premedication 1hr before treatment,which will be done in single visit.

After 1 hour, Pretreatment pain "pain after administration of analgesic or placebo" will be recorded using 0-10 numerical rating scale (NRS) .

Local anesthesia will, then, be done through inferior alveolar nerve block using 1.8 ml Mepivacaine.

The teeth will be isolated using rubber dam and access cavity will be prepared using #2 high-speed round bur.

The patients will be asked to rate their pain on the NRS. The degree of pain during access preparation and/or instrumentation will be recorded.

Success will be defined as no pain or mild pain during endodontic access preparation and/or instrumentation. Any pain more than no pain or mild pain will considered a failure.

The patients will be instructed to return after 2 days to complete the treatment procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aging between 18-50 years old.
2. Patients with mandibular molar with symptomatic irreversible pulpitis.
3. Systemically- healthy patients.
4. Patients who agree to attend for recall appointments and provide a written consent.

Exclusion Criteria:

1. Pregnant or lactating female patients.
2. Patients had allergies to any of test medications.
3. Patients had taken analgesics medication within the last 6 hours.
4. Moderate or severe marginal periodontitis i.e. pocket probe>3mm.
5. Non-restorable teeth, teeth with necrotic pulp, pulp polyp, tooth tender to percussion, root resorption or root canal calcification, periapical disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2021-01-09 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-07-11 (Actual)

PRIMARY OUTCOMES:
Success of mandibular inferior alveolar nerve block anesthesia during access and instrumentation. | During the treatment
  Will be recorded by 11 point NRS consisting of numbers from 0 through 10. 0: reading represents "no pain" 1-3 : readings represent "mild pain" 4-6 : readings represent "moderate pain" 7-10 : readings represent "severe pain" 0: reading represents "no pain" 1-3 : readings represent "mild pain" 4-6 : readings represent "moderate pain" 7-10 : readings represent "severe pain"

CONTACTS AND LOCATIONS:
Overall Officials: Alaa M. Morsi, Principal Investigator — Cairo University
Locations (1):
- Faculty of dentistry Cairo university, Giza, Non-US/Non-Canadian, Egypt

REFERENCES:
- [Background] Ianiro SR, Jeansonne BG, McNeal SF, Eleazer PD. The effect of preoperative acetaminophen or a combination of acetaminophen and Ibuprofen on the success of inferior alveolar nerve block for teeth with irreversible pulpitis. J Endod. 2007 Jan;33(1):11-4. doi: 10.1016/j.joen.2006.09.005. PMID 17185119
- [Background] Cohen HP, Cha BY, Spangberg LS. Endodontic anesthesia in mandibular molars: a clinical study. J Endod. 1993 Jul;19(7):370-3. doi: 10.1016/S0099-2399(06)81366-X. PMID 8245762
- [Background] Simpson M, Drum M, Nusstein J, Reader A, Beck M. Effect of combination of preoperative ibuprofen/acetaminophen on the success of the inferior alveolar nerve block in patients with symptomatic irreversible pulpitis. J Endod. 2011 May;37(5):593-7. doi: 10.1016/j.joen.2011.02.015. Epub 2011 Mar 22. PMID 21496654